CLINICAL TRIAL: NCT06039137
Title: The Effect of Switching the H1-antagonist Clemastine to Cetirizine in Premedication Regimens During Paclitaxel Treatment: 'The H1-SWITCH Study'
Brief Title: The Effect of Switching the H1-antagonist Clemastine to Cetirizine in Premedication Regimens During Paclitaxel Treatment
Acronym: H1-Switch
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Roelof W.F. van Leeuwen, Principal investigator, Erasmus Medical Center
Other Study IDs: METC 2022-0007
Record Dates: First submitted 2023-08-11; First posted 2023-09-15 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor
Keywords: Paclitaxel; Allergic reaction; HSR; Chemotherapy; Premedication; Cancer; Oncology
MeSH Terms: conditions — Hypersensitivity; Neoplasms | interventions — Cetirizine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clemastine group: Subjects receiving standard of care treatment with paclitaxel either as monotherapy or as part of a combination for any standard of care oncologic indication. Subjects received a paclitaxel premedication regimen containing dexamethasone 10 mg IV and clemastine 2 mg IV
  Interventions: Drug: Clemastine IV
- Cetirizine group: Subjects receiving standard of care treatment with paclitaxel either as monotherapy or as part of a combination for any standard of care oncologic indication. Subjects received a paclitaxel premedication regimen containing dexamethasone 10 mg IV and cetirizine 10 mg PO
  Interventions: Drug: Cetirizine

INTERVENTIONS:
Drug: Cetirizine — Subjects were treated with a paclitaxel premedication regimen which contained oral cetirizine instead of intravenous clemastine
  Groups: Cetirizine group
Drug: Clemastine IV — Subjects were treated with paclitaxel premedication containing clemastine 2 mg IV
  Groups: Clemastine group

SUMMARY:
In this study the effect of substituting clemastine IV to cetirizine PO on the occurence of hypersensitivity reactions during paclitaxel chemotherapy will be investigated.

DETAILED DESCRIPTION:
This is a single arm before-after study with a historic control cohort to evaluate the effect of a policy change (i.e. substitution of clemastine IV for cetirizine PO) regarding the premedication scheme on the incidence of HSR during paclitaxel based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Planned treatment with regular paclitaxel-based chemotherapy for any indication and with any dose

Exclusion Criteria:

* Prior treatment with a paclitaxel-based regimen;
* Inability to orally ingest cetirizine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors for whom paclitaxel-based chemotherapy is considered standard treatment will be eligible for this trial. Patients will be included from the outpatient population of the Erasmus MC in Rotterdam.
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Clinically relevant hypersensitivity reactions | During the first six cycles of paclitaxel treatment (the length of one cycle of paclitaxel treatment varies but is typically 7-21 days, depending on standard of care protocol).
  Hypersensitivity reactions grade 3 or higher according to CTCAE v4.03

SECONDARY OUTCOMES:
Hypersensitivity reactions | During the first six cycles of paclitaxel treatment (the length of one cycle of paclitaxel treatment varies but is typically 7-21 days, depending on standard of care protocol).
  Hypersensitivity reactions any grade according to CTCAE v4.03
The difference in the number of paclitaxel dosages until first occurrence of hypersensitivity reactions | During the first six cycles of paclitaxel treatment (the length of one cycle of paclitaxel treatment varies but is typically 7-21 days, depending on standard of care protocol).
  The difference in the number of paclitaxel dosages until first the occurrence of hypersensitivity reactions between the arms will be described.
The cumulative dose of paclitaxel (mg/m2) administered prior to the moment of hypersensitivity reaction | During the first six cycles of paclitaxel treatment (the length of one cycle of paclitaxel treatment varies but is typically 7-21 days, depending on standard of care protocol).
  The cumulative dose of paclitaxel (mg/m2) administered prior to the moment of occurrence of hypersensitivity reaction

CONTACTS AND LOCATIONS:
Overall Officials: Roelof van Leeuwen, PharmD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malmberg R, van Doorn L, Cox JM, Daloul A, Ettafahi H, Oomen-de Hoop E, Zietse M, Bos MEMM, Koch BCP, van Leeuwen RWF. Effect of Switching the Histamine-1 Receptor Antagonist Clemastine to Cetirizine in Paclitaxel Premedication Regimens: The H1-Switch Study. JCO Oncol Pract. 2024 Sep;20(9):1243-1251. doi: 10.1200/OP.24.00110. Epub 2024 Jun 7. PMID 38848522